CLINICAL TRIAL: NCT01103167
Title: The Association Between Body Composition and Biomarkers in Hemodialysis Patients
Brief Title: Body Composition Monitor in Hemodialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Gachon University Gil Medical Center IRB, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: korea_bcm_hd
Record Dates: First submitted 2010-04-09; First posted 2010-04-14 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: End Stage Renal Disease
Keywords: body composition; blood pressure; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: control of ultrafiltration — During the interventional period, dry weight of patients will be adjusted according to the results of body composition.

SUMMARY:
Control of volume status is a pivotal issue in haemodialysis therapy. Objective and practical management for maintaining normovolemia is needed.

The investigators hypothesized that intervention of volume status with the body composition monitor (BCM) may improved hemodynamic parameters and biomarkers in hemodialysis patients.

DETAILED DESCRIPTION:
The investigators will assess BCM in enrolled hemodialysis patients by 4 weeks for 16 weeks During the former 8-week intervention period, The investigators will adjust patients' volume status according to the results of BCM.

During the latter 8-week observational period, The investigators will evaluate the changes of patients' hemodynamic parameters and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 6-month or more stable hemodialysis patients
* 18 years or more
* less than 5% of changes of dry weight for last 3 months

Exclusion Criteria:

* pregnancy
* active malignancy
* cardiac pacemaker or defibrillator
* history of extremity amputation
* active infectious disease within 3 months
* admission history for complication related to hemodialysis within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
blood pressure | up to 16 weeks
  Systolic blood pressure, number of anti-hypertensive agents hypotensive episode

SECONDARY OUTCOMES:
biomarkers | up to 16 weeks
  C-reactive protein, interleukin-6, MMP-1, leptin, resistin, adiponectin, VEGF

CONTACTS AND LOCATIONS:
Overall Officials: Sejoong Kim, MD, PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Sejoong Kim, Incheon, South Korea